CLINICAL TRIAL: NCT02551497
Title: Double-Blind, Randomised, Placebo-Controlled, Parallel Group Study to Evaluate the Interaction Between a Drug and CNV1014802 in Healthy Subjects
Brief Title: Study to Evaluate the Interaction Between a Drug and CNV1014802 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1014802/102; 2015-001926-41 (EudraCT Number)
Record Dates: First submitted 2015-09-07; First posted 2015-09-16 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: volunteer drug interaction study
MeSH Terms: interventions — vixotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Other drug (Experimental): Other drug BID
  Interventions: Drug: CNV1014802
- placebo (Experimental): Placebo to match BID
  Interventions: Drug: CNV1014802

INTERVENTIONS:
Drug: CNV1014802

SUMMARY:
This is a double-blind, randomised, placebo-controlled 3 period study to evaluate the interaction between a drug and CNV1014802 in healthy male and female subjects. It is planned to enrol 36 subjects.

DETAILED DESCRIPTION:
This study was previously posted by Convergence Pharmaceuticals, Ltd., which has been acquired by Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, or non-pregnant, non-lactating healthy females either of non-child bearing potential, or taking an approved method of contraception for the duration of the study
* Age 18 to 55 years of age, inclusive
* Non-smoking subjects with body weight ≥45 kg
* Body mass index (BMI) of 18 to 32 kg/m2 (inclusive)
* Must be willing and able to communicate and participate in the whole study
* Must provide written informed consent
* Must agree to use an adequate method of contraception

Exclusion Criteria:

* Participation in a clinical research study within the previous 3 months
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee
* Subjects who have previously been enrolled in this study
* History of any drug or alcohol abuse in the past 2 years
* History of regular alcohol consumption within 6 months of the study (male subjects >21 units per week or female subjects >14 units per week; 1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
* Positive alcohol breath test
* Current smokers and those who have smoked within the last 6 months. A breath carbon monoxide reading of greater than 10 ppm at screening
* Females of childbearing potential who are pregnant or lactating (female subjects must have a negative urine pregnancy test at admission)
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
* Clinically significant abnormal biochemistry, haematology or urinalysis
* Positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* Positive genotyping test
* History of cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease as judged by the investigator
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than hormone replacement therapy [HRT]/hormonal contraception not containing ethinyl estradiol) or herbal remedies in the 14 days before IMP administration
* Significant medical history of fainting or vasovagal attacks
* History of uncontrolled or poorly controlled hypertension
* Semi-supine systolic BP <90 mmHg or >140 mmHg, or diastolic BP >100 mmHg after 3 assessments
* QTcB or QTcF of >450 msec in male subjects or >470 msec in females
* Presence or history of any clinically significant abnormality in vital signs or ECG
* Presence of any medical condition, which in the opinion of the investigator may interfere with the study procedures or compromise subject safety
* Medical history of clinically significant depression
* History of suicide attempt within 6 months prior to screening
* History of acute porphyria
* History of cardiac conduction disorders with the exception of 1st degree heart block
* Mentally or legally incapacitated
* Unwillingness or inability to follow the procedures outlined in the protocol, or to comply with study restrictions on smoking, concomitant medications and diet
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2016-08-16 (Actual); Study Completion 2016-08-26 (Actual)

PRIMARY OUTCOMES:
AUC(0-tau) of CNV1014802 and a drug | days 1-28
Cmax of CNV1014802 and a drug | 5 days
number of AEs | Days 16 to 21
heart rate | Days16-21
Blood pressure | Days16-21
ECG | Days 16-21
safety laboratory tests | Days 16-21

SECONDARY OUTCOMES:
CNV1014802 Tmax | days 1-28
CNV1014802 Ctrough | days 1-28

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Nottingham, United Kingdom